CLINICAL TRIAL: NCT02295280
Title: Metoclopramide and Diphenhydramine (MAD): A Cost Effective Treatment for Headache in Pregnancy When Acetaminophen Alone is Ineffective (MAD Headache Study)
Brief Title: A Cost Effective Treatment for Headache in Pregnancy When Acetaminophen Alone is Ineffective.
Acronym: MAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Dorothea Mostello, MD, MD, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15742
Record Dates: First submitted 2014-08-29; First posted 2014-11-20 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-02

CONDITIONS: Headache
Keywords: headache
MeSH Terms: conditions — Headache | interventions — Metoclopramide; Diphenhydramine; Codeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metoclopramide IV & Diphenhydramine IV (Active Comparator): Intravenous (IV) access will be obtained and administration of 10mg Metoclopramide IV and 25mg Diphenhydramine IV Group A
  Interventions: Drug: Metoclopramide; Drug: Diphenhydramine
- Codeine (Active Comparator): Group B (control group) will receive standard treatment consisting of a codeine 30mg tablet.
  Interventions: Drug: Codeine

INTERVENTIONS:
Drug: Metoclopramide — IV
  Other Names: metoclopramide, Reglan, Reglan ODT, Metozol ODT, Octamide,
  Arms: Metoclopramide IV & Diphenhydramine IV
Drug: Diphenhydramine — iv
  Other Names: Benadryl
  Arms: Metoclopramide IV & Diphenhydramine IV
Drug: Codeine — PO
  Arms: Codeine

SUMMARY:
To determine if the intravenous administration of Metoclopramide and diphenhydramine in combination can effectively treat headaches in pregnant patients in those refractory to acetaminophen when compared to codeine

DETAILED DESCRIPTION:
This is a randomized, controlled study based on prospective collection of data during the study subjects' hospital stays, questioning at 30 minutes and 1, 6, and 24 hours after administration, and a post-study questionnaire at 24 hours. Subjects who agree to participate in the study will have already tried a standard effective dose of acetaminophen (650 to 1000mg) without relief and are requesting further medication. Intravenous (IV) access will be obtained and administration of 10mg Metoclopramide IV and 25mg Diphenhydramine IV drawn up in the same syringe will be given to subjects randomized to Group A, while those randomized to Group B (control group) will receive standard treatment consisting of a codeine 30mg tablet. Each subject will be asked if they had relief or persistence/recurrence of symptoms at 30 minutes, 1 hour and 6 hours after initial receipt of study medications. An additional dose of 10 mg IV metoclopramide + 25 mg IV diphenhydramine or codeine 30 mg tablets would be given at one hour if the patient did not have adequate relief the first time. If headache does not subside or recurs after second dose, regular non protocol medicines may be administered upon doctor recommendation. Patients will again be asked about headache at 24 hours and asked to complete a questionnaire regarding tolerance of medication, any adverse reactions experienced, persistence/recurrence of headache after administration of study medication, timing of occurrence with regard to administration, requirements of a second dose of study medication or other use of headache or nausea medication not included in protocol, satisfaction or relief of headache on a Likert scale from 0 to 10 after administration of medication if given at 1 hr interval.

Randomization Subjects will be randomized to GROUP A or GROUP B. An order will be placed to the SMHC pharmacy for the respective Group and will send up the medication assigned. The pharmacy will know which medications are in Group A and which are in Group B. On the pharmacy order sheet, the research team will indicate which group each subject is randomized to. The pharmacy will supply the medications and one of the nurses on the 5th floor will administer them.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women age 16 or older, admitted to the hospital or treated in the triage unit at 14 weeks gestation or greater, with subjective symptoms of persistent headache despite 650-1000 mg acetaminophen taken more than one hour before administration of study medication.

Exclusion Criteria:

Treatment with another headache-aborting medication other than acetaminophen within 24 hours Allergy to metoclopramide, diphenhydramine, or codeine Systolic blood pressure >/= 140 Diastolic blood pressure >/= 90 History of brain tumor Active diagnosis of hyperemesis Acute asthma exacerbation at time of presentation Active labor

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothea Mostello, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective randomized, controlled trial at a single perinatal care center, conducted from December 2012 through September 2014 and approved by the IRB at Saint Louis University.
Period: Overall Study
Arm/Group | Metoclopramide IV & Diphenhydramine IV | Codeine
Started | 35 | 35
Completed | 35 | 34
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline demographic characteristics were similar between the two groups.
Groups:
- Metoclopramide IV & Diphenhydramine IV; Codeine: Normotensive pregnant women in the second or third trimester were randomized to receive either MAD intravenously (10 mg and 25 mg, respectively) or codeine (30 mg) for headache symptoms after 650-1000 mg of acetaminophen failed to relieve the headache.
- Total: Total of all reporting groups
Arm/Group | Metoclopramide IV & Diphenhydramine IV | Codeine | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 34 | 69
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 23 [21 to 25] | 23.5 [21 to 27] | 23 [21 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adequate Relief of Headache as a Measure of Efficacy
Description: Number of participants with reduction in pain scores six hours post administration by at least 2 on the pain score scale.
Time Frame: Primary outcome was six hours post administration
Population: Number in each arm with data at 6 hours who received either metoclopramide and diphenhydramine IV or codeine.
Measure: Count of Participants; unit: Participants
Groups:
- Metoclopramide IV & Diphenhydramine IV: Number of patients who received Metoclopramide & diphenhydramine IV
- Codeine: Number of patients who received codeine
Arm/Group | Metoclopramide IV & Diphenhydramine IV | Codeine
Number analyzed (Participants) | 34 | 32
Participants | 34 | 32
Statistical Analysis 1: Comparison: Metoclopramide IV & Diphenhydramine IV vs Codeine; A sample size calculation of 35 patients in each group was based on an estimated reduction in headache pain score by at least two points, with an a of 0.05 and power of 90%, which is similar to estimates reported in prior studies in non-pregnant patients and felt to be a clinically significant decrease. Statistical analyses were performed using chi-square, Fisher's exact test for categorical variables, the independent Student's t-test and Kolmogorov-Smirnov for continuous variables; Test type: Superiority; p = 0.14, Mann Whitney U test — Reduction in pain scores by at least 2 units six hours post administration; Mann Whitney U test used for analysis of this continuous variable as data were not normally distributed. Outcome was comparable at the 6-hour mark

ADVERSE EVENTS:
Time Frame: 24 hours
Description: No SAEs
Groups:
- Metoclopramide & Diphenhydramine: Participants received intravenous metoclopramine (10 mg) and diphenhydramine (25 mg), up to two doses of each medication.
- Codeine: Participants received oral 30 mg of oral codeine (up to two doses).
Arm/Group | Metoclopramide & Diphenhydramine | Codeine
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

LIMITATIONS AND CAVEATS:
One of the limitations of our study is that codeine was used as standard for comparison to the MAD regimen. This was due to poor patient enrollment with an earlier study design comparing MAD to placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No